CLINICAL TRIAL: NCT00612248
Title: Assessment of the Effectiveness of a Functional Splint for Osteoarthritis of the Trapeziometacarpal Joint on the Dominant Hand: A Randomized Controlled Study
Brief Title: Functional Splint for Osteoarthritis of the Trapeziometacarpal Joint
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Ana Claudia Gomes Carreira, UNIFESP - Universidade Federal de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIFESP0108; CEP1090/03
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Thumb; Splint; Pain; Function; Osteoarthritis of the trapeziometacarpal (TMC) joint
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SG (Experimental): Study group
  Interventions: Other: Splint
- CG (No Intervention): Control group

INTERVENTIONS:
Other: Splint — Patients in the study group received the splint on the day of the first evaluation and took it with them for use during activities of daily living and patients in the control group only used the splint during the evaluations
  Arms: SG

SUMMARY:
Forty participants were enrolled in a randomized, controlled clinical trial to evaluate the effectiveness of a functional thumb splint for trapeziometacarpal OA in the dominant hand.

DETAILED DESCRIPTION:
Treatment, Randomized, Single Blind, Placebo Control, Parallel Assignment, Efficacy Study

ELIGIBILITY:
Inclusion Criteria:

* clinical and radiological diagnosis of idiopathic Grade II and III OA of the TMC joint on the dominant hand;
* either gender;
* over 40 years of age;
* pain in the base of the thumb of the dominant hand greater than three and less than or equal to seven on the 0 to 10-cm visual analogue scale (VAS) for pain.

Exclusion Criteria:

* severe deformities of the dominant hand that did not allow gripping between the first, second and third fingers;
* deformities of distal interphalangeal joint;
* use of a splint on the thumb in the previous six months;
* surgery on the hand under study in the previous six months or scheduled in the upcoming six months;
* allergy to the splint material;
* incapacity to respond to the questionnaire and perform the tests;
* geographic inaccessibility;
* injections in the hand under study in the previous six months;
* other associated diseases such as carpal tunnel syndrome, fractures in the carpus, tendonitis, chronic inflammatory arthropathy;
* alterations in the use of anti-inflammatory medication and analgesics in the previous three months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | baseline (T0), after 45 days (T45), after 90 dias (T90) and after 180 dias (T180)

SECONDARY OUTCOMES:
Function (DASH) | baseline (T0), after 45 days (T45), after 90 dias (T90) and after 180 dias (T180)
Grip and pinch strength (dynamometer) | baseline (T0), after 45 days (T45), after 90 dias (T90) and after 180 dias (T180)
Dexterity (O'Connor test) | baseline (T0), after 45 days (T45), after 90 dias (T90) and after 180 dias (T180)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, MD, Study Chair — Federal University of São Paulo